CLINICAL TRIAL: NCT02887963
Title: Epidemiological Study of Iron Deficiency and Iron Deficiency Anemia Among Pregnant Women: A National Multicenter Survey in China
Brief Title: Epidemiological Study of Iron Deficiency and Iron Deficiency Anemia in Chinese Pregnant Women
Acronym: EIDACPW
Status: Completed | Type: Observational
Sponsor: West China Hospital (Other)
Collaborators: West China Second University Hospital (Other); Sichuan Provincial Hospital for Women and Children (Other); Panzhihua Central Hospital (Other); Chongqing Medical Center for Women and Children (Other); Obstetrics and Gynecology Hospital of Zhejiang University (Unknown); Xiamen Medical Center for Women and Children (Unknown); Wenzhou People's Hospital (Other); Suzhou Municipal Hospital (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Maternal and Child Health Hospital of Hubei Province (Other); The First Affiliated Hospital of Zhengzhou University (Other); First Affiliated Hospital of Guangxi Medical University (Other); Shanxi Provincial Maternity and Children's Hospital (Other); The Second Affiliated Hospital of Shanxi University of Traditional Chinese Medicine (Unknown); Yan'an University Affiliated Hospital (Other); Xinjiang Provincial Hospital for Women and Children (Unknown); Shengjing Hospital (Other); Dalian Maternity and Child Care Hospital (Other); Changchun Obstetrics and Gynecology Hospital (Unknown); The Fourth Affiliated Hospital of Harbin Medical University (Other); Beijing Obstetrics and Gynecology Hospital (Other); Tianjin Central Hospital of Gynecology Obstetrics (Other); The Fourth Hospital of Shijiazhuang (Other); Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Jing Tan, Chinese Evidence-based Medicine Centre, West China Hospital
Other Study IDs: IDA-China-2016
Record Dates: First submitted 2016-08-29; First posted 2016-09-02 (Estimated); Last update posted 2017-03-27 (Actual); Status verified 2017-03

CONDITIONS: Anemia, Iron-Deficiency
Keywords: Iron Deficiency; Iron Deficiency Anemia; Pregnant Women; Gestation; China; Epidemiology
MeSH Terms: conditions — Anemia, Iron-Deficiency; Iron Deficiencies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to know the prevalence of iron deficiency (ID) and iron deficiency anemia (IDA) among pregnant women in Chinese urban district at present, and to analyze the epidemiological characteristics of ID/IDA and influencing factors.

DETAILED DESCRIPTION:
This is a national large-scale multi-center cross-sectional survey aimed at investigating the epidemiology of iron deficiency (ID) and iron deficiency anemia (IDA) among Chinese pregnant women in the real world at present, which is anticipated to complete enrollment in two months. A total of 24 hospitals are selected from 6 regions (north, northeast, east, south, southwest, and northwest) of China by the method of multi-stage stratified sampling, each region with one tertiary teaching hospital and three general hospital or health care hospital for women and children. According to the sample size calculation formula combined with the feasibility and flexibility of study, 12000 eligible outpatient pregnant women are expected to be enrolled. Structured questionnaires, which are needed filled in both by patients and doctors, are used to collect participants' data, including basic demographic characteristics (age, occupation, educational level, family income, etc.), reproductive factors (menstrual history, times of pregnancy or parity, history of cesarean section, etc.), pre-pregnancy weight, pregnancy comorbidities and complications, laboratory test of blood routine and serum iron protein, use of iron supplements, diet and living habits during pregnancy, and others. The outcomes are defined by the recommendations on the guidelines for the diagnosis and treatment of Chinese iron deficiency and iron deficiency anemia during gestation period in 2014. All these data are requested to input the electronic data collecting (EDC) system in time and managed level-to-level, with Chinese Evidence-based Medicine Centre finally monitoring the quality of data. During the whole course, no intervention is given to the participants and thus will not have a negative effect on the health and rights of the participants.

ELIGIBILITY:
Inclusion Criteria:

* Receive outpatient service at selected hospitals for the first time during the survey period;
* Sign an informed consent form;
* At selected hospitals, establish registry of personal file for obstetric examination, or ensure regular follow-up.

Exclusion Criteria:

* Participate in any clinical trial of medicine or nutrition from 3 months before pregnancy till survey time.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Chinese pregnant women receiving outpatient service at selected hospitals
Sampling Method: Non-Probability Sample
Enrollment: 12000 (Actual)
Dates: Start 2016-09; Primary Completion 2016-11 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Iron Deficiency (ID) | two months
  serum ferritin concentration less than 20 μg/L
Iron Deficiency Anemia (IDA) | two months
  serum ferritin concentration less than 20 μg/L and hemoglobin less than 110 g/L

SECONDARY OUTCOMES:
Use of iron supplements | two months
  Iron agent type, dose and duration for preventing or treating ID/IDA

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese Evidence-based Medicine Centre, West China Hospital, Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided